CLINICAL TRIAL: NCT00162513
Title: Allogeneic Tumor Cell Vaccination in Patients With Chronic Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191199-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2006-09

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

INTERVENTIONS:
Biological: Allogeneic tumor cell vaccine

SUMMARY:
Donors with CM will be solicited from a waiting list of patients awaiting BMT from the waiting list of MUD searches.

Maximally matched donor will be searched for each eligible CML patient with a goal in mind to find other patients with CML that share both class I and class II determinants. Sharing of one class I II will be considered eligible for participation in the study. Peripheral blood and PBMC from the donors will be isolated, washed and irradiated.

The cells will be injected into the consenting patients intracutaneously at 2 weeks intervals for a total of 6 injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 55 consenting to participate in the study.
* Patients with documented CML with Philadelphia chromosome t (9:21)
* Patients with no HLA matched sibling.
* Patients eligible for BMT for who no matched unrelated donor can be identified after completion of an international donor search lasting for more than six months, or patients that have failed BMT.
* Patients with contra-indication to BMT.
* Patients refusing BMT.
* Patients who failed interferon alpha, ARAc and/or Glivec.

Exclusion Criteria:

* Patients requiring immunosuppressive therapy or corticosteroids.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-12

PRIMARY OUTCOMES:
Investigate the feasibility of allogeneic tumor cell vaccine for patients with resistant CML.

SECONDARY OUTCOMES:
To induce immunity against a putative bcr/abl peptide bound to MHC identical class I, II or preferably both.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel